CLINICAL TRIAL: NCT01249937
Title: Sub-tenon Triamcinolone Acetonide in Age-Related Macular Degeneration as Adjunct to Ranibizumab
Acronym: STAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Wai-Ching Lam, University Health Network-Toronto Western Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STARP2TWH
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-01

CONDITIONS: Wet Macular Degeneration
Keywords: Macular Degeneration; Age-related macular degeneration; Anti-inflammatory; Anti-vascular endothelial growth factor (Anti-VEGF); Lucentis; Ranibizumab; Kenalog; Triamcinolone Acetonide; Vision loss
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration; Vision Disorders | interventions — Ranibizumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Placebo Comparator): Ranibizumab is the current gold standard treatment for wet age-related macular degeneration. This intervention is approved by Health Canada, covered by OHIP (Ontario Health Insurance Plan) and used regularly by ophthalmologists in Canada. Participants will receive intravitreal injections of ranibizumab each month for up to 6 months, with ocular testing at each appointment as prescribed by the study protocol.
  Interventions: Drug: Ranibizumab
- Ranibizumab and Triamcinolone acetonide (Active Comparator): Recent research has discovered that persons with wet or dry ARMD show an immune response, as if the body is fighting off an infection. The body creates a complex immune response to the growth of blood vessels into the eye tissue, which triggers side effects. It is believed that preventing this inflammation can lead to greater visual gains and a need for fewer treatment injections.
  Animal studies have shown that Triamcinolone Acetonide, a corticosteroid (class of drugs that reduce inflammation) can prevent damage to vision from this inflammation. The hypothesis is that treatment with both Ranibizumab and Triamcinolone Acetonide will allow even greater vision improvements than Ranibizumab treatment alone for wet age-related macular degeneration.
  Interventions: Drug: Ranibizumab; Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Ranibizumab — Intra-vitreal injections of 0.5mg/0.05 mL dosage, injected at months 0, 1, and 2. For those requiring additional injections, patients will receive monthly treatment up to a maximum of 6 months total.
  Other Names: Lucentis
Drug: Triamcinolone Acetonide — Sub-tenon injection of 40mg/mL dosage at months 0 and 2 with follow up for a total of 6 months.
  Other Names: Kenalog
  Arms: Ranibizumab and Triamcinolone acetonide

SUMMARY:
In the Western World, Age Related Macular Degeneration (ARMD) is a leading cause of blindness. This disease was once thought to be a natural part of aging, but recent research has introduced effective treatments. ARMD is related to the body initiating an immune response in the eye, as if responding to an infection. Vision is impacted as ocular tissue becomes inflamed and new blood vessels form at the back of the eye, a process called angiogenesis. In the more severe wet form of ARMD, blood and fluid leak out of the vessels and impair the eye's structure and function. Many studies have shown that ranibizumab, a drug that stops the formation of new blood vessels (an anti-angiogenic agent) can delay damage to the eye and often restore vision. The investigators believe the best drug therapy will also stop the inflammation. Triamcinolone acetonide, a steroid drug, has shown the potential to effectively reduce inflammation in this application. The investigators aim to investigate if patients receiving a combination treatment of ranibizumab and triamcinolone acetonide improve their visual abilities more than those receiving just ranibizumab treatment alone. Secondarily, the investigators will also investigate how often patients receiving each drug therapy regime require re-treatment and how often they experience further vision loss.

DETAILED DESCRIPTION:
Age Related Macular Degeneration (ARMD or AMD) is the leading cause of blindness in North America. There are two types of ARMD: dry and wet. Both forms of ARMD cause a progressive loss of central vision, the part of your vision that allows you to read, drive and see images in sharp detail directly in front of you. The wet form is typically more severe and is characterized by the growth and leakage of small blood vessels into the choroid layer of the eye, or the back of the eye. These leaking blood vessels disrupt the structure and function of the eye, causing loss of vision, particularly the sharp vision created by the macula area of the eye.

Upon being accepted to the study, participants will be randomly divided into two groups. One group will receive both ranibizumab and triamcinolone acetonide injections and the other group will receive ranibizumab injections and a placebo treatment. To participants in this group, there will be the appearance of a second injection but no actual injection will take place. An individual not connected to the study will assign participants to a group based on a computer-generated system, giving participants at 50% chance of being placed in either group. During the study, participants will not know which group they are in, but will be able to know once the study is finished.

Participants will be asked to come in for an initial assessment to determine their starting visual abilities and medical history. On the next appointment, participants will receive the first treatment injections. They will be asked to come into the clinic every month for six (6) months total for treatment injections and testing. At each appointment, study investigators will take 3-D images of the retina (the back of the eye) using an Optical Coherence Tomography (OCT) imaging device, test eye pressure and determine if there are any signs of infection or inflammation from the injections. On months 1, 3 and 6 investigators will also test vision using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity charts, contrast sensitivity using a standard contrast sensitivity chart (The Pelli-Robson chart) and take images of the blood vessel growth using a coloured dye (fluorescein) to help see blood vessels. Before every treatment, anesthetic eye drops (proparacaine) will be applied to the eye so participants will not feel the injections. Participants will be given antibiotic eye drops (Zymar®) and will be asked to apply the drops 4 times a day for a few days after the injection to prevent infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with wet age-related macular degeneration (ARMD) with evidence of sub-foveal choroidal neo-vascularization (CNV)
* Patients greater than the age 18 years old (male or female)
* Visual acuity must be between 20/40 and 20/320 in the study eye.

Exclusion Criteria:

* Patients with CNV from causes other than ARMD
* Patients having intra-ocular surgery within past 3 months on study eye
* Patients with medically uncontrolled glaucoma
* Patients with prior vitreous/retinal surgery
* Patients with a history of past CNV treatment in study eye
* Patients with other ocular conditions causing vision loss that could confound the analysis of ARMD
* Individuals with a disability preventing accurate vision testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Gains in visual acuity | Baseline and months 1, 2, 3, 4, 5, and 6
  Gains in visual acuity will be assessed by comparing best corrected visual acuity at each follow up appointment by the standardized vision testing, early treatment diabetic retinopathy study (ETDRS) visual acuity test. The ETDRS visual acuity test was first developed to effectively evaluate visual changes following panretinal photocoagulation in patients with diabetic retinopathy. This method of measuring visual acuity was more accurate than previous methods, and thus has become the global standard, especially for clinical trials where it is essential to have utmost accuracy.

SECONDARY OUTCOMES:
Changes in intra-ocular pressure | Baseline and months 1, 2, 3, 4, 5 and 6
  To be measured by tonometry
Rates of re-treatment | Months 1, 2, 3, 4, 5 and 6
  To be measured by recording each drug administration date
Rate of vision loss | Baseline and months 1, 2, 3, 4, 5 and 6
  To be measured by ETDRS visual acuity testing and compared over the course of the study
Rate of cataract progression | Baseline and months 1, 2, 3, 4, 5, and 6
  Measured at each appointment with a slit lamp examination
• Changes in choroid vessel activity in lesion growth and activity at choroid | Baseline and months 1, 2, 3, 4, 5 and 6
  The changes in blood vessel lesion growth and activity will be measured by OCT (Ocular Coherence Tomography) and fundus fluoroscein angiography to assess choroidal neovascular leakage

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Ching Lam, MD, FRCSC, Principal Investigator — University Health Network, Toronto Western Hospital
Locations (1):
- University Health Network-Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Chaudhary V, Mao A, Hooper PL, Sheidow TG. Triamcinolone acetonide as adjunctive treatment to verteporfin in neovascular age-related macular degeneration: a prospective randomized trial. Ophthalmology. 2007 Dec;114(12):2183-9. doi: 10.1016/j.ophtha.2007.02.013. PMID 18054638